CLINICAL TRIAL: NCT01151436
Title: Global Management of Facial Rejuvenation With a New Range of Hyaluronic Acid Dermal Fillers - Investigator and Subject Satisfaction
Brief Title: Global Management of Facial Rejuvenation With a New Range of Hyaluronic Acid Dermal Fillers
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.CIP.29089; 2009-018163-28 (EudraCT Number)
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2012-05

CONDITIONS: Facial Wrinkles
Keywords: Facial wrinkle correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hyaluronic acid (Experimental)
  Interventions: Device: hyaluronic acid dermal fillers

INTERVENTIONS:
Device: hyaluronic acid dermal fillers — 1 injection per indication and 1 touch-up injection if necessary
  Other Names: Facial wrinkles

SUMMARY:
The aim of this study is to assess performance and tolerance as well as investigator and subject satisfaction linked to the global management of facial rejuvenation with a new range of hyaluronic acid dermal fillers.

DETAILED DESCRIPTION:
The range of fillers tested in this study includes 5 different hyaluronic acid dermal fillers: Emervel Touch, Emervel Classic, Emervel Deep, Emervel Volume and Emervel Lips.

The study will last 6 month.

Injections will be performed at baseline. If necessary, the investigator will perform touch-up injections at the following visit (3 weeks later).

Investigator and subject satisfaction will be collected through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Seeking tissue augmentation treatment on the face,
* Presenting a score of 3 (Moderately deep wrinkle)or 4 (Deep wrinkle) on the Lemperle Rating Scale (LRS) of both nasolabial folds.

Exclusion Criteria:

* At risk in term of precautions, warnings and contra-indication referred in the package insert of the study devices,
* Who underwent previous injection of permanent filler in the injected area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe KESTEMONT, Principal Investigator — Investigational site Nice France
Locations (5):
- France (3):
  - Galderma investigational site, Arras
  - Galderma investigational site, Nice
  - Galderma investigational site, Paris
- Germany (2):
  - Galderma investigational site, Berlin
  - Galderma investigational site, Darmstadt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyaluronic Acid
Started | 77
Completed | 76
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 4
Region of Enrollment [Number; unit: participants]
  France | 47
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Full Face Global Aesthetic Improvement
Description: Global aesthetic improvement scale score from baseline:
  -1: worse 0: no change
  1. improved
  2. much improved
  3. very much improved
Time Frame: 3 weeks after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 77
units on a scale | 2.5 (0.6)

2. Secondary Outcome: NASOLABIAL FOLDS SEVERITY ASSESSMENT
Description: Severity scored on Lemperle Rating Scale:
  0: no wrinkles
  1. just perceptible wrinkle
  2. shallow wrinkle
  3. moderately deep wrinkle
  4. deep wrinkle, well-defined edges
  5. very deep wrinkle redundant fold
Time Frame: baseline
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wrinkle
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 73
Number analyzed (wrinkle) | 146
units on a scale | 3.4 (0.5)

3. Primary Outcome: Full Face Global Aesthetic Improvement
Description: as for outcome 1
Time Frame: 3 months after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 75
units on a scale | 2.4 (0.6)

4. Primary Outcome: Full Face Global Aesthetic Improvement
Description: as for outcome 1
Time Frame: 6 months after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 76
units on a scale | 1.8 (0.9)

5. Secondary Outcome: NASOLABIAL FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 weeks after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wrinkle
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 73
Number analyzed (wrinkle) | 146
units on a scale | 1.4 (0.9)

6. Secondary Outcome: NASOLABIAL FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 months after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wrinkle
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 71
Number analyzed (wrinkle) | 142
units on a scale | 1.6 (0.8)

7. Secondary Outcome: NASOLABIAL FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 6 months after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: wrinkle
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 72
Number analyzed (wrinkle) | 144
units on a scale | 2 (1)

8. Secondary Outcome: PERIORBITAL LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: baseline
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 31
Number analyzed (WRINKLE) | 62
units on a scale | 2.9 (1)

9. Secondary Outcome: PERIORBITAL LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 weeks after last injection
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 31
Number analyzed (WRINKLE) | 62
units on a scale | 1.7 (1)

10. Secondary Outcome: PERIORBITAL LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 31
Number analyzed (WRINKLE) | 62
units on a scale | 1.8 (1)

11. Secondary Outcome: PERIORBITAL LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 6 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 31
Number analyzed (WRINKLE) | 62
units on a scale | 2.1 (1.2)

12. Secondary Outcome: MARIONETTE LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: BASELINE
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLES
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 68
Number analyzed (WRINKLES) | 136
units on a scale | 3.1 (1)

13. Secondary Outcome: MARIONETTE LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 WEEKS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 68
Number analyzed (WRINKLE) | 136
units on a scale | 1.4 (1)

14. Secondary Outcome: MARIONETTE LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 MONTHS AFTER LAST INJECTION
Population: ININTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 66
Number analyzed (WRINKLE) | 132
units on a scale | 1.6 (1)

15. Secondary Outcome: MARIONETTE LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 6 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 67
Number analyzed (WRINKLE) | 134
units on a scale | 2 (1.1)

16. Secondary Outcome: UPPER LIP LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: BASELINE
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 44
Number analyzed (WRINKLE) | 44
units on a scale | 3.1 (1)

17. Secondary Outcome: UPPER LIP LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 WEEKS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 44
Number analyzed (WRINKLE) | 44
units on a scale | 1.5 (0.9)

18. Secondary Outcome: UPPER LIP LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 44
Number analyzed (WRINKLE) | 44
units on a scale | 1.7 (0.9)

19. Secondary Outcome: UPPER LIP LINES SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 6 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 43
Number analyzed (WRINKLE) | 43
units on a scale | 2.1 (0.9)

20. Secondary Outcome: CHEEK FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: BASELINE
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 28
Number analyzed (WRINKLE) | 55
units on a scale | 2.4 (0.6)

21. Secondary Outcome: CHEEK FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 WEEKS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 28
Number analyzed (WRINKLE) | 55
units on a scale | 1.3 (0.6)

22. Secondary Outcome: CHEEK FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 3 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 27
Number analyzed (WRINKLE) | 53
units on a scale | 1.4 (0.6)

23. Secondary Outcome: CHEEK FOLDS SEVERITY ASSESSMENT
Description: as for outcome 2
Time Frame: 6 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: WRINKLE
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 27
Number analyzed (WRINKLE) | 53
units on a scale | 1.8 (0.8)

24. Secondary Outcome: LIP ENHANCEMENT ASSESSMENT
Description: Lip fullness grading scale score:
  0: very thin lip
  1. thin lip
  2. moderately thick lip
  3. thick lip
  4. full lip
Time Frame: baseline
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: number of lips (upper or lower)
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 44
Number analyzed (number of lips (upper or lower)) | 71
units on a scale | 1.2 (0.7)

25. Secondary Outcome: LIP ENHANCEMENT ASSESSMENT
Description: Lip fullness grading scale score:
  0: very thin lip
  1. thin lip
  2. moderately thick lip
  3. thick lip
  4. full lip
Time Frame: 3 WEEKS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: number of lips (upper or lower)
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 44
Number analyzed (number of lips (upper or lower)) | 71
units on a scale | 2.3 (0.8)

26. Secondary Outcome: LIP ENHANCEMENT ASSESSMENT
Description: Lip fullness grading scale score:
  0: very thin lip
  1. thin lip
  2. moderately thick lip
  3. thick lip
  4. full lip
Time Frame: 3 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: number of lips (upper or lower)
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 43
Number analyzed (number of lips (upper or lower)) | 70
units on a scale | 2.2 (0.9)

27. Secondary Outcome: LIP ENHANCEMENT ASSESSMENT
Description: Lip fullness grading scale score:
  0: very thin lip
  1. thin lip
  2. moderately thick lip
  3. thick lip
  4. full lip
Time Frame: 6 MONTHS AFTER LAST INJECTION
Population: INTENT TO TREAT ON OBSERVED POPULATION (NO REPLACEMENT OF MISSING VALUE)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: number of lips (upper or lower)
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 43
Number analyzed (number of lips (upper or lower)) | 70
units on a scale | 2 (0.9)

ADVERSE EVENTS:
Time Frame: During the study period (maximum of 24 weeks)
Arm/Group | Hyaluronic Acid
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 5/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronic Acid (N=77)
NASOPHARYNGITIS (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor to review and approval at least 2 months prior to the date of intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.